CLINICAL TRIAL: NCT04119440
Title: A Two-center, Randomized, Double-blind, Placebo-controlled, Phase Ib Study to Assess the Safety, Tolerability and Immunogenicity of Two Ascending Doses of the Candidate Vaccine MVA-MERS-S_DF-1 in Healthy Study Subjects
Brief Title: Safety and Immunogenicity of the Candidate Vaccine MVA-MERS-S_DF-1 Against MERS
Acronym: MVA-MERS-S
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); IDT Biologika Dessau.Rossau (Unknown); German Center for Infection Research (Other); CR2O (Unknown); Erasmus Medical Center (Other); Monipol Deutschland GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEPI-MVA-MERS-S-Phase1b
Record Dates: First submitted 2019-10-06; First posted 2019-10-08 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: MERS (Middle East Respiratory Syndrome)
Keywords: MERS-CoV; CEPI; viral vector vaccine
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded with an open-label run-in Phase (Part A) Part A: Open-label Part B: Double-blind
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose (Experimental): Vaccination with 2x10^7 PFU MVA-MERS-S_DF1. Vaccinations will be administered at days 0, 28 or 56, and 336.
  Interventions: Biological: MVA-MERS-S_DF1 - Low Dose
- High Dose (Experimental): Vaccination with 2x10^8 PFU MVA-MERS-S_DF1. Vaccinations will be administered at days 0, 28 or 56, and 336.
  Interventions: Biological: MVA-MERS-S_DF1 - High Dose
- Placebo (Placebo Comparator): Injection with placebo. Injections will be administered at days 0, 28 or 56, and 336.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MVA-MERS-S_DF1 - Low Dose — Administrations of the low dose via the intramuscular route
  Arms: Low Dose
Biological: MVA-MERS-S_DF1 - High Dose — Administrations of the high dose via the intramuscular route
  Arms: High Dose
Other: Placebo — Administrations of placebo via the intramuscular route
  Arms: Placebo

SUMMARY:
The study will be a two center, randomized, double blind, placebo controlled study of the MVA MERS S_DF-1 candidate delivered by i.m. injection. To evaluate the MERS-S-specific antibody responses and safety profile induced by the two dosage levels of MVA-MERS-S_DF-1 the data will be compared to a placebo control group.

DETAILED DESCRIPTION:
This will be a Phase Ib, two-center study in approximately 160 healthy adults aged 18-55 years

The study is separated in two parts:

Part A:

The study starts with a single center open-label run-in phase of two dose levels (cohort 1 "low dose": 2x10^7 PFU, cohort 2 "high dose": 2x10^8 PFU) in 10 healthy subjects. 5 subjects will be allocated to each dose cohort and will receive immunization on day 0 and day 28.

Part B:

Two-center, randomized, double-blind, placebo-controlled, dose-finding study. This part is a double-blinded trial in approximately 150 healthy subjects. Subjects will be allocated to two different dose cohorts and a placebo cohort; each receiving three vaccine injections.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent form.
2. Healthy male and female subjects aged 18-55 years.
3. No clinically significant acute health problems as determined from medical history and physical examination at screening visit.
4. Body mass index 18.5 - 30.0 kg/m2 and weight > 50 kg at screening.
5. Non-pregnant, non-lactating female with negative pregnancy test.
6. Males and females who agree to comply with the applicable contraceptive requirements of the protocol.

Exclusion Criteria:

1. Receipt of any vaccine from 2 weeks prior to each trial vac-cination (4 weeks for live vaccines) to 3 weeks after each trial vaccination.
2. Receipt of vaccination against MERS or MVA immunizations.in the medical history.
3. Known allergy to the components of the MVA-MERS-S_DF-1 vaccine product.
4. Evidence in the subject's medical history or in the medical examination that might influence either the safety of the subject or the absorption, distribution, metabolism or excretion of the investigational product.
5. Any confirmed or suspected immunosuppressive or immuno-deficient condition, cytotoxic therapy in the previous 5 years, and/or diabetes.
6. Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events associated with MVA-MERS-S_DF-1. | day 1, 14, 29, 42, 56, 84, 168, 336, 364
  Safety and reactogenicity will be assesssed by observation, questionaire and diary. Changes from baseline for safety laboratory measures will be monitored. Occurence of SAE will be collected throughout the entire study duration.
Frequency and severity of local injection site reactogenicity signs and symptoms | day 1, 14, 29, 42, 84, 336

SECONDARY OUTCOMES:
Immunogenicity | day 0, 14, 28, 42, 56, 70, 84, 168, 336, 364 (dependent on vaccination scheme)
  Magnitude of MERS-S-specific antibody re-sponses (ELISA and neutralization assays) monitored in a centralized approved laboratory

CONTACTS AND LOCATIONS:
Locations (2):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Erasmus Medical Centre, Rotterdam, Rotterdam, Netherlands

REFERENCES:
- [Derived] Raadsen MP, Dahlke C, Fathi A, Hardtke S, Kluver M, Krahling V, Gerresheim GK, Mayer L, Mykytyn AZ, Weskamm LM, Zoran T, van Gorp ECM, Sutter G, Becker S, Haagmans BL, Addo MM; MVA-MERS-S_DF-1 Study group. Safety, immunogenicity, and optimal dosing of a modified vaccinia Ankara-based vaccine against MERS-CoV in healthy adults: a phase 1b, double-blind, randomised placebo-controlled clinical trial. Lancet Infect Dis. 2025 Feb;25(2):231-242. doi: 10.1016/S1473-3099(24)00423-7. Epub 2024 Oct 7. PMID 39389076